CLINICAL TRIAL: NCT05374577
Title: Pulmonary Vascular Dysfunction as a Cause of Persistent Exertional Dyspnea After COVID-19 (PulmVasC)- A Multicenter, Prospective Cohort/Observational Study
Brief Title: Pulmonary Vascular Dysfunction as a Cause of Persistent Exertional Dyspnea After Coronavirus Disease (COVID-19)
Acronym: PulmVasC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: KKS-300
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a suspected diagnosis of post/long-COVID-19: Patients with a suspected post-COVID-19 syndrome or a long-COVID-19 syndrome at least 3 months after severe acute respiratory syndrome coronavirus(CoV) type 2 (SARS-CoV-2) infection (symptomatic or asymptomatic)
  Interventions: Other: pulmonary vascular dysfunction
- Patients without post/long-COVID-19 Syndrome: Patients at least 3 months after a SARS-CoV-2 infection (symptomatic or asymptomatic) without post/long-COVID-19.
  Interventions: Other: pulmonary vascular function

INTERVENTIONS:
Other: pulmonary vascular dysfunction — Right ventricular function determined by echocardiography at rest and during exercise (non-invasive estimation of ventilation-perfusion mismatch), systemic endothelial function, left heart function, and plasma levels of vasoactive biomarkers compared with clinical parameters of dyspnea and exercise capacity. Further examinations will be performed in patients with still unclear cause of persistent shortness of breath after 3 months of follow-up (subgroup RHC)
  Groups: Patients with a suspected diagnosis of post/long-COVID-19
Other: pulmonary vascular function — Right ventricular function determined by echocardiography at rest and during exercise (non-invasive estimation of ventilation-perfusion mismatch), systemic endothelial function, and plasma levels of vasoactive biomarkers compared with clinical parameters of dyspnea and exercise capacity.
  Groups: Patients without post/long-COVID-19 Syndrome

SUMMARY:
To identify pulmonary vascular disease in post/long-COVID-19 patients as a cause of dyspnea/exercise limitation and to differentiate it from other causes of dyspnea

DETAILED DESCRIPTION:
The aim is to identify pulmonary vascular disease in post/long-COVID-19 patients as a cause of dyspnea/exercise limitation and to differentiate it from other causes of dyspnea (muscular, left cardiac, psychological, deconditioning-related causes) by investigating ventilation-perfusion (V/Q) mismatch and (exercise-induced) pulmonary hypertension (PH) or right heart dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, patients with a suspected diagnosis of post/long-COVID-19 syndrome who present to our pneumology or infectious disease outpatient clinic or corresponding ward from the start of the study and whose SARS-CoV-2 infection was diagnosed at least 3 and not longer than 18 months prior to presentation
* Patients at least 3 and not longer than 18 months after a SARS-CoV-2 infection without post/long-COVID-19 syndrome who present to our post-infection outpatient clinic for follow-up

Exclusion Criteria:

* Patients who refuse to participate in the study
* Severe underlying chronic pulmonary, cardiac, or systemic disease (e.g., Chronic obstructive pulmonary disease (COPD), severe heart failure, neuromuscular disease) that was diagnosed prior to acute COVID-19 disease and whose progression appears likely as the cause of dyspnea
* Other non pneumologic causes of dyspnea (e.g., hemoglobin < 100 g/L)
* Unstable or acute disease (e.g., acute infection, acute renal failure, acute coronary syndrome)
* Inability to perform spiroergometry, including transient orthopedic problems, contraindications to central venous and arterial catheter placement (e.g., severe bleeding tendency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a post-COVID-19 syndrome or a long-COVID-19 syndrome at least 3 months after SARS-CoV-2 infection (symptomatic or asymptomatic); Patients at least 3 months after a SARS-CoV-2 infection (symptomatic or asymptomatic) without post/long-COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of gas exchange under different inhaled oxygen concentrations | At the time of presentation (on day 1)
  Non-invasive estimation of ventilation/perfusion (V/Q) mismatch
Spiroergometric capacity- maximal oxygen uptake (VO2max; ml/min/kg) | At the time of presentation (on day 1)
  Determination of exercise capacity by cardiopulmonary exercise testing (CPET)
Echocardiographic right heart parameters - pulmonary arterial systolic pressure (PASP; mmHg) | At the time of presentation (on day 1)
  Echocardiographic determination of right heart parameters under rest and during exercise
Echocardiographic right heart parameters - Tricuspid annular plane systolic excursion (TAPSE; mm) | At the time of presentation (on day 1)
  Echocardiographic determination of right heart parameters under rest and during exercise
Echocardiographic right heart parameters - right ventricular (RV) end-ventricular volume (EDV; ml) | At the time of presentation (on day 1)
  Echocardiographic determination of right heart parameters under rest and during exercise
Echocardiographic right heart - right volume (RV) end-systolic volume (ESV; ml) | At the time of presentation (on day 1)
  Echocardiographic determination of right heart parameters under rest and during exercise
Echocardiographic right heart - right ventricular longitudinal global strain (%) | At the time of presentation (on day 1)
  Echocardiographic determination of right heart parameters under rest and during exercise
Dyspnoea Index | At the time of presentation (on day 1)
  Determination of dyspnea and functional capacity a questionaire measure of shortness of breath for determining exertion levels
Invasive hemodynamics - pulmonary vascular resistance (PVR; WU) | At the time of presentation (on day 1)
  Invasive measurement of pulmonary hemodynamics by right heart catheterization (RHC subgroup)
Invasive hemodynamics - cardiac Index (CI; l/min/m2) | At the time of presentation (on day 1)
  Invasive measurement of pulmonary hemodynamics by right heart catheterization (RHC subgroup)

SECONDARY OUTCOMES:
Left heart parameters - (E/e' ratio) | At the time of presentation (on day 1)
  Determination of left heart parameters during rest and exercise
Left heart parameters - left ventricular ejection fraction (%) | At the time of presentation (on day 1)
  Determination of left heart parameters during rest and exercise
Pulmonary vascular function | At the time of presentation (on day 1)
  Increase of echocardiographically estimated systolic pulmonary arterial pressure during inhalation of hypoxic gas
Airway Impedance | At the time of presentation (on day 1)
  Determination of airway impedance by oscillometry
Peripheral blood mononuclear cells | At the time of presentation (on day 1)
  Determination of characteristics of peripheral immune cells by fluorescence activated cell sorter (FACS) and functional assays
Shunt measurement | At the time of presentation (on day 1)
  Shunt measurement by contrast-enhanced echocardiography (optional)
Ventilation/Perfusion mismatch | At the time of presentation (on day 1)
  Determination of V/Q mismatch using the gold standard multiple inert gas elimination technique (MIGET) (only in RHC subgroup)
Static and dynamic lung function parameters - vital capacity (VC; L) | At the time of presentation (on day 1)
  Determination of lung function by body plethysmography at rest
Static and dynamic lung function parameters - forced expiratory volume in 1 s (FEV1; L) | At the time of presentation (on day 1)
  Determination of lung function by body plethysmography at rest
Static and dynamic lung function parameters - diffusion capacity (DLCO; %) | At the time of presentation (on day 1)
  Determination of lung function by body plethysmography at rest
Static and dynamic lung function parameters - diffusion coefficient (DLCO/VA; %) | At the time of presentation (on day 1)
  Determination of lung function by body plethysmography at rest

CONTACTS AND LOCATIONS:
Overall Officials: Natascha Sommer, PD, Principal Investigator — Cardiopulmonary Institute (CPI), University of Giessen and Marburg Lung Center (UGMLC)
Locations (1):
- Natascha Sommer, Giessen, Germany

REFERENCES:
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Gierhardt M, Pak O, Walmrath D, Seeger W, Grimminger F, Ghofrani HA, Weissmann N, Hecker M, Sommer N. Impairment of hypoxic pulmonary vasoconstriction in acute respiratory distress syndrome. Eur Respir Rev. 2021 Sep 15;30(161):210059. doi: 10.1183/16000617.0059-2021. Print 2021 Sep 30. PMID 34526314
- [Background] Nuzzi V, Castrichini M, Collini V, Roman-Pognuz E, Di Bella S, Luzzati R, Berlot G, Confalonieri M, Merlo M, Stolfo D, Sinagra G. Impaired Right Ventricular Longitudinal Strain Without Pulmonary Hypertension in Patients Who Have Recovered From COVID-19. Circ Cardiovasc Imaging. 2021 Apr;14(4):e012166. doi: 10.1161/CIRCIMAGING.120.012166. Epub 2021 Apr 8. No abstract available. PMID 33827250
- [Background] Rossi R, Coppi F, Monopoli DE, Sgura FA, Arrotti S, Boriani G. Pulmonary arterial hypertension and right ventricular systolic dysfunction in COVID-19 survivors. Cardiol J. 2022;29(1):163-165. doi: 10.5603/CJ.a2021.0159. Epub 2021 Dec 13. No abstract available. PMID 34897638
- [Background] Reichenberger F, Voswinckel R, Schulz R, Mensch O, Ghofrani HA, Olschewski H, Seeger W. Noninvasive detection of early pulmonary vascular dysfunction in scleroderma. Respir Med. 2009 Nov;103(11):1713-8. doi: 10.1016/j.rmed.2009.05.004. Epub 2009 Jun 3. PMID 19497725
- [Background] Kjaergaard S, Rees S, Malczynski J, Nielsen JA, Thorgaard P, Toft E, Andreassen S. Non-invasive estimation of shunt and ventilation-perfusion mismatch. Intensive Care Med. 2003 May;29(5):727-34. doi: 10.1007/s00134-003-1708-0. Epub 2003 Apr 16. PMID 12698242
- [Background] Thomsen LP, Karbing DS, Smith BW, Murley D, Weinreich UM, Kjaergaard S, Toft E, Thorgaard P, Andreassen S, Rees SE. Clinical refinement of the automatic lung parameter estimator (ALPE). J Clin Monit Comput. 2013 Jun;27(3):341-50. doi: 10.1007/s10877-013-9442-9. Epub 2013 Feb 21. PMID 23430364
- [Background] Trinkmann F, Benck U, Halder J, Semmelweis A, Saur J, Borggrefe M, Akin I, Kaden JJ. Automated Noninvasive Central Blood Pressure Measurements by Oscillometric Radial Pulse Wave Analysis: Results of the MEASURE-cBP Validation Studies. Am J Hypertens. 2021 Apr 20;34(4):383-393. doi: 10.1093/ajh/hpaa174. PMID 33140085
- [Background] Winkler J, Hagert-Winkler A, Wirtz H, Hoheisel G. [Modern impulse oscillometry in the spectrum of pulmonary function testing methods]. Pneumologie. 2009 Aug;63(8):461-9. doi: 10.1055/s-0029-1214938. Epub 2009 Aug 7. German. PMID 19670105
- [Background] Wagner PD. The multiple inert gas elimination technique (MIGET). Intensive Care Med. 2008 Jun;34(6):994-1001. doi: 10.1007/s00134-008-1108-6. Epub 2008 Apr 18. PMID 18421437
- [Background] Shah W, Hillman T, Playford ED, Hishmeh L. Managing the long term effects of covid-19: summary of NICE, SIGN, and RCGP rapid guideline. BMJ. 2021 Jan 22;372:n136. doi: 10.1136/bmj.n136. No abstract available. PMID 33483331
- [Background] Sonnweber T, Sahanic S, Pizzini A, Luger A, Schwabl C, Sonnweber B, Kurz K, Koppelstatter S, Haschka D, Petzer V, Boehm A, Aichner M, Tymoszuk P, Lener D, Theurl M, Lorsbach-Kohler A, Tancevski A, Schapfl A, Schaber M, Hilbe R, Nairz M, Puchner B, Huttenberger D, Tschurtschenthaler C, Asshoff M, Peer A, Hartig F, Bellmann R, Joannidis M, Gollmann-Tepekoylu C, Holfeld J, Feuchtner G, Egger A, Hoermann G, Schroll A, Fritsche G, Wildner S, Bellmann-Weiler R, Kirchmair R, Helbok R, Prosch H, Rieder D, Trajanoski Z, Kronenberg F, Woll E, Weiss G, Widmann G, Loffler-Ragg J, Tancevski I. Cardiopulmonary recovery after COVID-19: an observational prospective multicentre trial. Eur Respir J. 2021 Apr 29;57(4):2003481. doi: 10.1183/13993003.03481-2020. Print 2021 Apr. PMID 33303539
- [Background] Augustin M, Schommers P, Stecher M, Dewald F, Gieselmann L, Gruell H, Horn C, Vanshylla K, Cristanziano VD, Osebold L, Roventa M, Riaz T, Tschernoster N, Altmueller J, Rose L, Salomon S, Priesner V, Luers JC, Albus C, Rosenkranz S, Gathof B, Fatkenheuer G, Hallek M, Klein F, Suarez I, Lehmann C. Post-COVID syndrome in non-hospitalised patients with COVID-19: a longitudinal prospective cohort study. Lancet Reg Health Eur. 2021 Jul;6:100122. doi: 10.1016/j.lanepe.2021.100122. Epub 2021 May 18. PMID 34027514